CLINICAL TRIAL: NCT06532773
Title: Mindfulness Intervention for Sleep Disturbance and Symptom Management in Hematologic Cancer Patients During and After Inpatient Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00115799; K08CA283026 (NIH)
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-07

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nite2Day+ (Experimental): During inpatient treatment, Nite2Day+ will be delivered via a self-paced mobile app. Participants will use the app to access: 1) mindfulness meditations (e.g., Body Scan, 3-Minute Mini-Meditation) from Mindfulness Based Therapy for Insomnia (MBTI); 2) brief, 3-5 minute sleep education videos (i.e., 3-P Model of Insomnia, sleep hygiene, sleep drive, circadian rhythm) specifically tailored to the inpatient setting; and 3) brief, 3-5 minute videos teaching behavioral strategies (e.g., stimulus control, daytime activity, light exposure, communication with medical team) to improve sleep quality in the hospital. After inpatient treatment, Nite2Day+ will deliver a six session (45-60 minutes), therapist-led, Zoom protocol. Participants will learn new mindfulness-based sleep strategies (e.g., sleep consolidation, sleep reconditioning), meditations (e.g., Sitting Meditation), and behavioral symptom coping skills.
  Interventions: Behavioral: Nite2Day+
- Usual Care (No Intervention): Participants will receive written materials describing free services (e.g., legal and financial assistance, counseling) available through the Duke Cancer Patient Support Program.

INTERVENTIONS:
Behavioral: Nite2Day+ — Mindfulness-based sleep strategies and cognitive-behavioral symptom coping skills.
  Other Names: Mindfulness Based Therapy for Insomnia; Cognitive Behavioral Symptom Coping Skills
  Arms: Nite2Day+

SUMMARY:
People with hematologic cancer often have sleep disturbance and symptoms of fatigue, stress, and pain. This study is being done to test a mindfulness intervention for sleep disturbance and symptom management in patients with hematologic cancer during and after inpatient treatment (Nite2Day+). Participants will complete a baseline survey online, using a mobile application, or paper/pencil. Once the baseline survey is complete, participants will be randomized (like a flip of a coin) to receive Nite2Day+ or Standard Care. Nite2Day+ will include activities during and after inpatient treatment. During inpatient treatment, participants will use a mobile app to access: 1) mindfulness meditations, 2) brief sleep education videos, and 3) brief videos teaching strategies to improve sleep quality in the hospital. After inpatient treatment, participants will complete 6, videoconference sessions (45-60 minutes) with a trained therapist to learn mindfulness and behavioral coping strategies to self-manage nighttime sleep disturbance and daytime symptoms of fatigue, stress, and pain. Three follow-up surveys will occur at hospital discharge, and approximately 8, and 12 weeks after hospital discharge. Participants randomized to Nite2Day+ will be given the option to complete an exit interview to provide feedback on the Nite2Day+ program. Participants randomized to Standard Care will only complete the four surveys. All participants will continue to receive their usual medical care. The total study duration is about 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients, >18 years old
2. Initial or recurrent diagnosis of acute myeloid leukemia, acute lymphoblastic leukemia, Non-Hodgkin's lymphoma, multiple myeloma, or myelodysplastic syndrome
3. at least 7 days of hospitalization for treatment (e.g., chemotherapy, CAR-T immunotherapy)
4. 8 or greater on the Insomnia Severity Index with timeframe adjusted to be "past 7 days"
5. Ability to speak and read English, and intact hearing and vision

Exclusion Criteria:

1. Reported or suspected cognitive impairment, confirmed via Folstein Mini-Mental Status Exam <25
2. Serious psychiatric (e.g., schizophrenia, suicidal intent) or medical condition (e.g., seizure disorder, narcolepsy) indicated by medical chart, oncologist, or other provider
3. Expected survival of <6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility as measured by study accrual | 24 months of study recruitment
  Treatment feasibility will be shown by meeting targeted study accrual (N = 60 in 24 months).
Feasibility as measured by study attrition | Baseline (0 weeks), Discharge (4 weeks), Post-Intervention (13 weeks), 1-month post-intervention (17 weeks)
  Treatment feasibility will be shown by no more than 25% study attrition.
Feasibility as measured by adherence | Baseline (0 weeks), Discharge (4 weeks), Post-Intervention (13 weeks), 1-month post-intervention (17 weeks)
  Adherence will be indicated by at least 75% of study sessions and assessments completed.
Acceptability as measured by the Client Satisfaction Questionnaire (CSQ) | Baseline (0 weeks), Discharge (4 weeks), Post-Intervention (13 weeks), 1-month post-intervention (17 weeks)
  Acceptability will be indicated by at least 80% of the participants reporting satisfaction with the protocol on the CSQ. Items are rated on a 4-point scale from 1 (low) to 4 (high) and averaged to obtain an acceptability score ranging from 1 to 4, with higher scores indicating higher acceptability.
Engagement as measured by Nite2Day+ app and skills use | Baseline (0 weeks), Discharge (4 weeks), Post-Intervention (13 weeks), 1-month post-intervention (17 weeks)
  Engagement will be indicated by Nite2Day+ app log-in and skills practice at least 2 times per week.
Change in insomnia symptoms | Baseline (0 weeks), Discharge (4 weeks), Post-Intervention (13 weeks), 1-month post-intervention (17 weeks)
  Insomnia symptoms will be measured using the 7-item Insomnia Symptom Index (ISI). Items are summed to yield a total score ranging from 0 to 28, with higher scores indicating worse insomnia symptoms.

SECONDARY OUTCOMES:
Change in fatigue | Baseline (0 weeks), Discharge (4 weeks), Post-Intervention (13 weeks), 1-month post-intervention (17 weeks)
  Fatigue symptoms will be assessed using the 8-item PROMIS Fatigue Short Form. A raw score is calculated by summing all 8 items, yielding a total raw score that ranges from 8 to 40. The total raw score is then translated to a T-score, which is a standardized score with a mean of 50 and a standard deviation of 10. Higher T-scores indicated higher fatigue.
Change in depressive symptoms | Baseline (0 weeks), Discharge (4 weeks), Post-Intervention (13 weeks), 1-month post-intervention (17 weeks)
  Depressive symptoms will be assessed using the 8-item PROMIS Depression Short Form. A raw score is calculated by summing all 8 items, yielding a total raw score that ranges from 8 to 40. The total raw score is then translated to a T-score, which is a standardized score with a mean of 50 and a standard deviation of 10. Higher T-scores indicate higher worse depressive symptoms.
Change in anxiety symptoms | Baseline (0 weeks), Discharge (4 weeks), Post-Intervention (13 weeks), 1-month post-intervention (17 weeks)
  Anxiety symptoms will be assessed using the 8-item PROMIS Anxiety Short Form. A raw score is calculated by summing all 8 items, yielding a total raw score that ranges from 8 to 40. The total raw score is then translated to a T-score, which is a standardized score with a mean of 50 and a standard deviation of 10. Higher T-scores indicate worse anxiety symptoms.
Change in pain severity | Baseline (0 weeks), Discharge (4 weeks), Post-Intervention (13 weeks), 1-month post-intervention (17 weeks)
  Pain severity will be assessed using the 11-item Brief Pain Inventory-Short Form (BPI-SF). The BPI-SF consists of 4 items assessing pain severity, including worst, least, average, and current pain in the past week. Responses range from 0 (no pain) to 10 (pain as bad as you can imagine); items are averaged for a composite score that ranges from 0 to 10 with higher scores indicating high pain severity.
Change in pain interference | Baseline (0 weeks), Discharge (4 weeks), Post-Intervention (13 weeks), 1-month post-intervention (17 weeks)
  Pain interference will be assessed using the 11-item Brief Pain Inventory-Short Form (BPI-SF). The BPI-SF consists of 7 items assessing the degree to which pain has interfered with patients' daily activities in the past week. Responses range from 0 (does not interfere) to 10 (completely interferes); items are averaged for a composite score that ranges from 0 to 10 with higher scores indicating high pain interference.
Change in mindfulness | Baseline (0 weeks), Discharge (4 weeks), Post-Intervention (13 weeks), 1-month post-intervention (17 weeks)
  Mindfulness will be assessed using the 10-item Cognitive and Affective Mindfulness Scale - Revised. Participants will be asked to rate their level of mindfulness across two domains (cognitive and affective) using a 4-point response scale ranging from 1 (rarely/not at all) to 4 (almost always). Items are summed to yield a total score, with higher scores reflecting greater mindfulness.
Change in self-efficacy for symptom management | Baseline (0 weeks), Discharge (4 weeks), Post-Intervention (13 weeks), 1-month post-intervention (17 weeks)
  Self-efficacy for symptom management will be assessed using the 8-item PROMIS Self-Efficacy for Managing Chronic Conditions - Managing Symptoms Scale. Participants will rate their confidence in managing their symptoms using a 5-point response scale from 1 (I am not at all confident) to 5 (I am very confident). Items are summed and converted to a T-score, which is a standardized score with a mean of 50 and a standard deviation of 10. Higher T-scores indicate better self-efficacy for symptom management.

CONTACTS AND LOCATIONS:
Locations (1):
- 2400 Pratt Street, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No